CLINICAL TRIAL: NCT01037998
Title: Phase II Trial of Adding UFUR to Non-small-cell Lung Cancer Patients Treated With Iressa
Brief Title: UFUR (Tegafur/Uracil) Plus Iressa in Non-small-cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Yuh-Min Chen, MD, PhD, Associate Professor, Chest Department
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 94-09-03
Record Dates: First submitted 2008-05-27; First posted 2009-12-23 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2009-12

CONDITIONS: Non-Small-Cell Lung Cancer
Keywords: adenocarcinoma; non-small-cell lung cancer; gefitinib; UFUR
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Adenocarcinoma | interventions — Tegafur; Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Iressa 250 mg daily treatment plus UFUR twice daily treatment
  Interventions: Drug: UFUR and Iressa
- B (No Intervention): Gefitinib 250 mg daily treatment

INTERVENTIONS:
Drug: UFUR and Iressa — Iressa 250 mg daily plus UFUR 1# bid
  Other Names: UFUR
  Arms: A

SUMMARY:
Iressa [epidermal growth factor tyrosine kinase inhibitor (EGFR-TKI)] has been reported to activity against Non-small-cell Lung Cancer (NSCLC) failed previous chemotherapy. UFUR was found to have anti-angiogenesis effect when long term treatment was given. Combination of EGFR-TKI and anti-angiogenesis agents is a novel treatment.

DETAILED DESCRIPTION:
Iressa is a selective epidermal growth factor receptor tyrosine kinase inhibitor (EGFR-TKI). It is an orally active agent for advanced non-small-cell lung cancer (NSCLC) in those who have failed a previous platinum-based regimen and taxane treatment. UFUR (Tegafur/Uracil) is effective agent against chemo-naïve NSCLC. It has anti-angiogenesis effect when used as long-term low dose treatment.

Present phase II randomized clinical trial is designed to answer whether or not adding an oral anti-angiogenesis agent (UFUR), that has low toxicity profiles when long term use, to EGFR-TKI (Iressa) could increase patients survival and response rate.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytological diagnosis of NSCLC who failed previous platinum-based and taxanes chemotherapy.
* No prior radiotherapy on measurable lesion(s).
* Performance status of 0 to 3 on the Zubrod scale. (Reference 1)
* Clinically measurable disease, defined as bidimensionally measurable lesions with clearly defined margins on x-ray, scan, or physical examination. Lesions serving as measurable disease must be at least 1 cm by 1 cm, as defined by CT scan, MRI, or chest x-ray.
* Informed consent from patient.
* Males or females 18 years of age or older.
* If female: childbearing potential either terminated by surgery, radiation, or menopause, or attenuated by use of an approved contraceptive method (intrauterine contraceptive device [IUD], birth control pills, or barrier device) during and for three months after trial.

Exclusion Criteria:

* Active infection (at the discretion of the investigator).
* Inadequate liver function (total bilirubin >1.5 times above normal range); alanine transaminase (ALT) and aspartate transaminase (AST) greater than 5 times normal.
* Inadequate renal function (creatinine >2.0 mg/dL).
* Breast feeding.
* Second primary malignancy (except in situ carcinoma of the cervix or adequately treated basal cell carcinoma of the skin)
* Concomitant myelosuppressive radiotherapy, chemotherapy, hormonal therapy, or immunotherapy will not be allowed except as for palliative radiation to non-measurable lesion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2005-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To assess and compared the 6-month survival rate of these two arms of treatment. | 6 months

SECONDARY OUTCOMES:
To assess and compared the progression-free survival, overall survival, the response rate, and the toxicity profiles of these two arms of treatment. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yuh-Min Chen, MD, PhD., Principal Investigator — Chest Department, Taipei VGH
Locations (1):
- Taipei VGH, Taipei, Taiwan